CLINICAL TRIAL: NCT02881632
Title: Pneumacare SLP Validation in Infants and in Clinical Bronchiolitis: Validation of Structured Light Plethysmography (SLP) in Healthy Infants and in Infants With Clinical Bronchiolitis
Brief Title: Pneumacare SLP Validation in Infants and in Clinical Bronchiolitis
Status: Completed | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Collaborators: Pneumacare Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 836
Record Dates: First submitted 2016-04-28; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy infants aged 0-2: Healthy infants aged 0-2 year with no respiratory diseases to provide a reference values. A structured light pattern (Structured Light Plethysmography (SLP) - Pneumscan) will be projected onto the chest and abdominal wall and the movement of this pattern as the patient breathes will be recorded for 2 min. The total period of testing per session should take approximately 30 minutes per person.
  Interventions: Device: Structured Light Plethysmography (SLP) - Pneumscan
- Infants aged 0-1 with Bronchiolitis: Infants admitted to hospital within last 24hrs (AVB participants only). A structured light pattern (Structured Light Plethysmography (SLP) - Pneumscan) will be projected onto the chest and abdominal wall and the movement of this pattern as the patient breathes will be recorded for 2 min. The total period of testing per session should take approximately 30 minutes per person
  Interventions: Device: Structured Light Plethysmography (SLP) - Pneumscan

INTERVENTIONS:
Device: Structured Light Plethysmography (SLP) - Pneumscan — Both healthy infants and bronchiolitis infants will have their chest movements monitored using Structured Light Plethysmography (SLP) performed by a device (Thora-3 Di) using a projector and two cameras. A light pattern of black and white squares is projected on the child's chest and the cameras record how the shape of this pattern changes with breathing. A computer converts this information to show how the child's chest moves during breathing.

SUMMARY:
A cohort observational study to characterise baseline Structured Light Plethysmography (SLP) outputs in infants with bronchiolitis and examine response to treatment using the Thora3DiTM

DETAILED DESCRIPTION:
Viral illness, particularly chest infection causing breathing difficulty in infants and children is the commonest reason for admission to hospital. At present, there are no objective measurements of the degree of breathing difficulty.

This is because current objective tests of breathing difficulty requires the patient to cooperate and actively perform the tests. This is not possible in babies and very challenging in young children. SLP is a noncontact, effort independent technique for measuring the rate of breathing, the amount of chest expansion and the relative contribution of chest and abdomen to the work of breathing. Measuring these parameters which are known to vary with increasing breathing difficulty will allow us to make objective assessments of breathing difficulty. This study proposes to validate this technique in babies aged 02 years who are healthy and in babies with clinical viral bronchiolitis. The Investigators intend to demonstrate that the technique is feasible in this young age group and that the investigators will be able to demonstrate clinically valid differences between normal and ill babies and also demonstrate measurable differences with the evolution of the clinical illness.

ELIGIBILITY:
Inclusion Criteria

* Aged between 0 and 1 years
* Doctor diagnosis of AVB
* Admitted to hospital within last 24hrs (AVB participants only)
* Or healthy term infant aged up to 2yrs with no current respiratory illness

Exclusion Criteria:

* Patients with significant co morbidities resulting in clinical instability (assessed by the clinician at screening only):
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in the study
* Parents unable to consent/comply with trial protocol
* An inpatient for over 24hrs (AVB patients only)

Ages: 1 Minute to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants aged 0-2 years and Infants aged 0-1 years with Bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Difference in SLP measurements between infants. | Measured upto 7 days
  Difference in SLP measurements between infants. SLP provides a measure of the chest and abdominal movement (Respiratory effort) of the subjects, the movement signal will be used to quantify clinically relevant tidal breathing parameters such as timing indices: Ti (Time of inspiration), Te ( Time of expiration) and Ttot (Ti+Te). Parameters will be quantified for each recorded SLP signal (averaged) from each infant, and then used to compare between infants with bronchiolitis and healthy babies.

SECONDARY OUTCOMES:
Changes in SLP measurements in infants during their clinical course. | Measured upto 7 days
  Changes in SLP measurements in infants during their clinical course in hospital. SLP provides a measure of the chest and abdominal movement (Respiratory effort) of the subjects, the movement signal will be used to quantify clinically relevant tidal breathing parameters such as timing indices: Ti (Time of inspiration), Te ( Time of expiration) and Ttot (Ti+Te). For each subject SLP was recorded on a daily basis, this will allow the comparison between the parameters within subject to check the progression of the disease with time
Changes in SLP measurements in infants given additional breathing support. | Measured upto 7 days
  Changes in SLP measurements in infants during their clinical course in hospital who are given additional breathing support. SLP provides a measure of the chest and abdominal movement (Respiratory effort) of the subjects, the movement signal will be used to quantify clinically relevant tidal breathing parameters such as timing indices: Ti (Time of inspiration), Te ( Time of expiration) and Ttot (Ti+Te). For each subject SLP was recorded on a daily basis, this will allow the comparison between the parameters within subject to check the progression of the disease with time.

CONTACTS AND LOCATIONS:
Overall Officials: John Alexander, Principal Investigator — UHNM
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No